CLINICAL TRIAL: NCT01245608
Title: Fixed-dose Combination Therapy (PolyPill) in Prevention of Cardiovascular Disease in Middle-aged and Elderly Iranians - Focus on Liver-Related Variables.
Brief Title: Prevention of Cardiovascular Disease Using a Single PolyPill in an Urban Population - Focus on Liver-Related Variables.
Acronym: PolyIran-L
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Golestan University of Medical sciences (Other); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 90-03-37-15582
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2018-02

CONDITIONS: Cardiovascular Diseases
Keywords: Atorvastatin; Aspirin; nonalcoholic steatohepatitis; nonalcoholic fatty liver disease; antihypertensive agents
MeSH Terms: conditions — Cardiovascular Diseases; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Polypill (Experimental): Single daily dose of PolyPill and 6-monthly visits
  Interventions: Drug: Polypill
- Control (No Intervention): Only 6-monthly visits

INTERVENTIONS:
Drug: Polypill — Polypill taken once daily for 5 years. Each pill contains acetylsalicylic acid 81 mg, atorvastatin 20 mg, hydrochlorothiazide 12.5 mg, valsartan 40 mg
  Other Names: PolyPill 4-2
  Arms: Polypill

SUMMARY:
The primary purpose of this study is to determine the effects of a fixed dose combination of valsartan, hydrochlorothiazide, atorvastatin and aspirin (PolyPill) on prevention of cardiovascular events in adults older than 50.

Various liver-related variables will also be recorded which will allow studying the effects of PolyPill on the liver and the effect of liver diseases such as nonalcoholic steatohepatitis on cardiovascular events and the protective effect of PolyPill.

DETAILED DESCRIPTION:
2400 subjects will be randomly selected from participants of the Golestan Cohort Study (GCS) who are living in Gonbad and are over 50 years old. These subjects will be randomized to either receive PolyPill or no treatment.

Those agreeing to the study will undergo additional measurements (in addition to the baseline measurements performed in the GCS) including liver-related tests such as liver enzyme levels, abdominal ultrasonography and liver stiffness measurement. Some additional tests such as color doppler ultrasonography of carotid vessels will also be performed.

Subjects in the PolyPill arm who have no contraindication for the components of the pill will receive a single daily dose of PolyPill for 5 years.

ELIGIBILITY:
Inclusion Criteria:

- Being enrolled in Golestan Cohort Study

Exclusion Criteria:

* Debilitating disease causing inability to comply
* Contraindications to any of the components of PolyPill
* Not consenting to the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Major Cardiovascular Events | 5 years
  The first occurrence of hospitalization for acute coronary syndrome (non-fatal myocardial infarction and unstable angina), fatal myocardial infarction, sudden death, new-onset heart failure, coronary artery revascularization procedures and stroke (fatal or non-fatal).

SECONDARY OUTCOMES:
Side effects | 5 years
  questionnaire
Changes in liver enzyme levels | 5 years
  AST, ALT
Changes in liver stiffness | 5 years
  As measured by fibroscan
Compliance | 5 years
  Pill count
Fat deposition | 5 years
  Visceral Adipose Tissue thickness (VAT), Subcutaneous Adipose Tissue thickness (SAT) and carotid intima-media thickness (IMT)
All-cause Mortality | 5 years
  Yearly follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Reza Malekzadeh, M.D., Study Chair — Tehran University of Medical Sciences; Shahin Merat, M.D., Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Golestan Cohort Center, Gonbad, Golestan Province, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pourshams A, Khademi H, Malekshah AF, Islami F, Nouraei M, Sadjadi AR, Jafari E, Rakhshani N, Salahi R, Semnani S, Kamangar F, Abnet CC, Ponder B, Day N, Dawsey SM, Boffetta P, Malekzadeh R. Cohort Profile: The Golestan Cohort Study--a prospective study of oesophageal cancer in northern Iran. Int J Epidemiol. 2010 Feb;39(1):52-9. doi: 10.1093/ije/dyp161. Epub 2009 Mar 30. No abstract available. PMID 19332502
- [Background] Ostovaneh MR, Poustchi H, Hemming K, Marjani H, Pourshams A, Nateghi A, Majed M, Navabakhsh B, Khoshnia M, Jaafari E, Mohammadifard N, Malekzadeh F, Merat S, Sadeghi M, Naemi M, Etemadi A, Thomas GN, Sarrafzadegan N, Cheng KK, Marshall T, Malekzadeh R. Polypill for the prevention of cardiovascular disease (PolyIran): study design and rationale for a pragmatic cluster randomized controlled trial. Eur J Prev Cardiol. 2015 Dec;22(12):1609-17. doi: 10.1177/2047487314550803. Epub 2014 Sep 17. PMID 25230980
- [Derived] Merat S, Jafari E, Radmard AR, Khoshnia M, Sharafkhah M, Nateghi Baygi A, Marshall T, Shiravi Khuzani A, Cheng KK, Poustchi H, Malekzadeh R. Polypill for prevention of cardiovascular diseases with focus on non-alcoholic steatohepatitis: the PolyIran-Liver trial. Eur Heart J. 2022 Jun 1;43(21):2023-2033. doi: 10.1093/eurheartj/ehab919. PMID 35048107
- [Derived] Merat S, Poustchi H, Hemming K, Jafari E, Radmard AR, Nateghi A, Shiravi Khuzani A, Khoshnia M, Marshall T, Malekzadeh R. PolyPill for Prevention of Cardiovascular Disease in an Urban Iranian Population with Special Focus on Nonalcoholic Steatohepatitis: A Pragmatic Randomized Controlled Trial within a Cohort (PolyIran - Liver) - Study Protocol. Arch Iran Med. 2015 Aug;18(8):515-23. PMID 26265520